CLINICAL TRIAL: NCT06179433
Title: Outcome of Regenerative Endodontic Procedure in Comparison to Nonsurgical Root Canal Treatment for the Management of Necrotic Mature Molar Teeth With Periapical Lesions - A Randomized Controlled Trial
Brief Title: Outcome of Regenerative Endodontic Procedure and Root Canal Treatment for the Management of Apical Periodontitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dr.Jigyasa Duhan
Record Dates: First submitted 2023-12-12; First posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Apical Periodontitis
Keywords: regenerative endodontics, root canal treatment
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- root canal treatment (Experimental): Two-visit root canal treatment will be performed.
  Interventions: Procedure: Root canal treatment
- REP with I-PRF (Active Comparator): The first appointment will be performed similar to the conventional RCT group. in the second appointment, i-PRF will be prepared by collecting venous blood and centrifugate at 700rpm for 3 minutes. i-PRF will be injected into canal followed by a bioceramic material.
  Interventions: Procedure: Regenerative endodontic procedure
- REP with blood clot (Active Comparator): The first appointment will be performed similar to the conventional RCT group. In the second appointment, after anesthetizing with 3% mepivacine, the canals will be re-entered and irrigated well with 17% EDTA. Bleeding will be induced by inserting sterile #25 K-file into the 2-3 mm beyond the apical foramen into periapical tissues.
  Interventions: Procedure: Regenerative endodontic procedure

INTERVENTIONS:
Procedure: Root canal treatment — Two-visit root canal treatment will be performed.
  Arms: root canal treatment
Procedure: Regenerative endodontic procedure — Regenerative endodontic procedure with i-PRF and blood clot induction will be performed.
  Arms: REP with I-PRF; REP with blood clot

SUMMARY:
Background Root canal therapy is the primary treatment of choice for necrotic mature teeth with periapical lesions (PRLs), which does not restore the tooth's vitality. Provided that injectable platelet-rich fibrin (i-PRF) has shown promising results in regenerative medicine as a novel platelet concentration, the purpose of this study is to ascertain whether i-PRF, as opposed to blood clot (BC), can serve as a biological scaffold, thereby expanding the indications for regenerative endodontic procedures (REPs) in mature teeth.

Novelty There is no study available that has evaluated the outcome of REP in the necrotic mature mandibular molars with periapical lesions. Furthermore, the efficacy of novel i-PRF as a scaffold in REPs remains to be explored.

Objectives To evaluate and compare the outcome of REPs in comparison to conventional RCT in necrotic mature molars with PRLs and to evaluate the efficacy of i-PRF and BC in REP as a scaffold. Secondary objective is to evaluate pain for first postoperative week and subjective responses to pulp sensibility tests at 12 months follow-up.

Method 120 patients presenting with necrotic pulp and periapical lesions will be randomly allotted to one of the three groups - REP using i-PRF or BC or RCT group. Comparative evaluation of outcome of REP and RCT will be performed at 12-months follow-up.

DETAILED DESCRIPTION:
Regenerative endodontic procedures (REPs) are biologically based procedures used to replace damaged structures such as dentin and root structures, as well as pulp-dentin complex cells (4, 5). Majority of studies have focused on treating immature necrotic teeth with the REP approach in order to preserve root development and regenerate functional pulp tissue (6-9). REPs have recently been proposed as an alternative approach to treating necrotic mature permanent teeth with apical periodontitis due to their promising results (10-12). However, it did face a few challenges, including fewer stem cells, narrower apical foramina for induction of blood and stem cell migration, and difficulty disinfecting the root completely (11).

The most common scaffold for revascularization involves creation of blood clot (BC) by inducing bleeding from the periapical tissue using an endodontic file. However, blood clots are a meagre source of growth factors, and the precise method required to control the rate and volume of bleeding is still uncertain (13-15). Second-generation platelet concentrate, or platelet-rich fibrin (PRF), is a type of natural autologous fibrin matrix containing trapped leukocytes and platelets to ensure a sustained release of cytokines and growth factors. However, their applicability is restricted because of its solid nature. The development of a liquid form of PRF (injectable PRF) in 2016 was made possible by the use of gentle or low speed centrifugation, which has benefits for bone, periodontal cartilage, and pulp tissue regeneration (16,17). After application, injectable PRF (i-PRF) gradually changes into a growth factor-rich PRF clot that releases growth factors steadily over the course of 10 to 14 days (16).

To the best of our knowledge, no study has been conducted that utilized i-PRF as a scaffold for REPs in mature teeth. Therefore, the aim of this trial is to evaluate and compare the efficacy of i-PRF and blood clot as scaffolds in REPs in comparison to nonsurgical root canal treatment in necrotic mature molars with periapical lesions (PRLs).

ELIGIBILITY:
Inclusion Criteria:

1. Consenting healthy adults with age range of 18- 40 years
2. Patient presenting with atleast one permanent mandibular molar with necrotic pulp (negative response to sensibility testing by cold and electric pulp test).
3. Radiographic evidence of periapical radiolucency of strictly endodontic origin score ≥3 according to the classification of Ørstavik et al (diagnosis of asymptomatic apical periodontitis or chronic apical abscess) with lesion size ≤ 5mm

Exclusion Criteria:

* Non-restorable teeth or tooth with severe coronal defect where rubber dam isolation is not possible
* Teeth with root fractures or pathological root resorptions
* Teeth with endodontic- periodontal communications
* Patients with generalized chronic periodontitis or periodontal pocket more than 3 mm
* Teeth with previous root canal treatment
* Severe root canal curvatures
* Pregnant or lactating women
* Patients with a history of systemic diseases and/or receiving medications that affect healing or blood coagulation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
clinical and radiographic success | 12 month follow-up.
  Clinical and radiographic success of REPs in comparison to conventional RCT in necrotic mature molars with PRLs

SECONDARY OUTCOMES:
postoperative pain | 1 week
  Postoperative pain at first week after procedure
Pulp sensibility response | 6 and 12 months
  Subjective response to pulp sensibility test

CONTACTS AND LOCATIONS:
Overall Officials: jigyasa 1 duhan, MDS, Principal Investigator — PGIDS
Locations (1):
- postgraduate Institute of Dental sciences, Rohtak, Haryana, India